CLINICAL TRIAL: NCT05318287
Title: Walk With Me (WWM) for Perinatal Grief
Brief Title: Walk With Me for Perinatal Grief
Acronym: PeriGrief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MH126788
Record Dates: First submitted 2022-02-01; First posted 2022-04-08 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Grief; Traumatic Stress; Usability
MeSH Terms: interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PeriGrief (Experimental): A brief four-module intervention delivered via computer or mobile device. Modules utilize mindfulness and cognitive behavioral therapy strategies to reduce distress following perinatal loss.
  Interventions: Behavioral: Walk with Me

INTERVENTIONS:
Behavioral: Walk with Me — Walk with Me is a perinatal grief mobile application to provide supportive care to bereaved parents. The application includes modules to guide bereaved parents through strategies to help support them through their grieving.

SUMMARY:
This research will contribute to therapeutic technology to support bereaved parents who have experienced a perinatal loss. The proposed mobile application would accomplish this objective by providing a series of therapeutic modules to provide parents with tools to normalize their grief and additional coping skills to support the grieving process.

DETAILED DESCRIPTION:
The investigators will develop grief processing and healing activities for bereaved parents, via an iterative formative development process with stakeholder input. The investigators will embed the core intervention components in administrative, provider, and client interfaces which will comprise the prototype Walk with Me (WWM) intervention.

The investigators will evaluate its feasibility and initial efficacy of WWM in a within-subjects pre-post design study. The investigators will provide the mobile-based provider component for use by health care professionals (HCPs) who work in the partner hospital. HCPs will have access to training videos and bereaved parent content. After training, the HCPs will recruit 52 bereaved parents.

HCPs will obtain consent from bereaved parents who express interest in the study to share their contact information with the research team. Parents who wish to participate will provide consent for their own participation in the study. After consent, parents will complete the baseline survey via the Qualtrics online assessment form and then be provided download access to the WWM prototype. At 4 and 8 weeks, parents will be administered post-treatment surveys. This design will allow the investigators to evaluate baseline to follow-up change in the proposed study outcomes and acceptability of the prototype WWM program.

Baseline and post-treatment surveys will measure bereaved parents traumatic stress, grief intensity, grief, grief management self-efficacy, and care experiences. The post-survey questionnaire will contain measures of usability, as well as any difficulties experienced or problems made worse. Demographics will be collected at the baseline assessment. Project staff will follow-up with parents as needed to encourage survey completion in a timely manner.

ELIGIBILITY:
Inclusions Criteria

Focus Groups and Usability Testing (Bereaved Parents)

* Experienced a perinatal loss
* Have had at least 6 months pass since experiencing the most recent loss
* Age 15 and older

Efficacy Study (Bereaved Parents)

* Bereaved parent who has experienced a perinatal loss within the last two weeks * Age 15 and older
* Have access to technology to view WWM content

Exclusion Criteria

* Non-English speakers are excluded. The WWM program will first be developed in English and its feasibility established.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille C Cioffi, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PeriGrief
Started | 52
Completed | 44
Not Completed | 8
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 6
  White | 36
  More than one race | 3
  Unknown or Not Reported | 3
Relationship Status [Count of Participants; unit: Participants]
  Single, dating | 1
  Married or domestic partner | 45
  Partnered in a serious relationship | 5
  Divorced or separated | 1
Number of times pregnant [Count of Participants; unit: Participants]
  1 | 13
  2 | 18
  3 | 12
  4 | 4
  5 or more | 5
Type of loss experienced - Chemical Pregnancy (i.e., loss before the 5th week) [Count of Participants; unit: Participants] | 4
Type of loss experienced - Miscarriage in the first trimester [Count of Participants; unit: Participants] | 21
Type of loss experienced - Neonatal loss [Count of Participants; unit: Participants] | 7
Type of loss experienced - Stillbirth [Count of Participants; unit: Participants] | 11
Type of loss experienced - Termination due to fetal abnormality/viability [Count of Participants; unit: Participants] | 4
Type of loss experienced - Tubal or ectopic pregnancy [Count of Participants; unit: Participants] | 1
Type of loss experienced - Tubal or ectopic pregnancy [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Traumatic Stress - Intrusion Subscale
Description: Impact of Event Scale-Revised (IES-R) includes 22 items on the past 7 days that represent symptoms of distress self-rated on a five-point scale: 0 indicates that the symptom occurs "not at all"; 1, "a little bit"; 2, "moderately"; 3, "quite a bit"; and 4, "extremely." Participants will be instructed to relate the IES-R items specifically to the loss of their child. Three scale scores are computed including intrusions (8 items), avoidance (8 items) and hyperarousal (6 items). Each subscale ranges from 0 to 4 with higher scores indicating greater levels of distress/trauma.
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: There were 52 participants with pretest data, 48 with 4-weeks data, and 44 is 8-weeks data. Trajectories were estimated using maximum likelihood and thus, any participant with at least one data point was included in the analyses. Thus, all 52 participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 2.17 (0.92)
  4-weeks: number analyzed (Participants) | 48
  4-weeks | 1.93 (0.90)
  8-weeks: number analyzed (Participants) | 44
  8-weeks | 1.32 (1.01)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .083, t-test, 2 sided; Slope = -0.05, Standard Error of Mean 0.03

2. Primary Outcome: Traumatic Stress - Avoidance Subscale
Description: Impact of Event Scale-Revised includes 22 items on the past 7 days that represent symptoms of distress self-rated on a five-point scale: 0 indicates that the symptom occurs "not at all"; 1, "a little bit"; 2, "moderately"; 3, "quite a bit"; and 4, "extremely." Participants will be instructed to relate the IES-R items specifically to the loss of their child. Three scale scores are computed including intrusions (8 items), avoidance (8 items) and hyperarousal (6 items). Each subscale ranges from 0 to 4 with higher scores indicating greater levels of distress/trauma.
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 1.61 (0.93)
  4-weeks: number analyzed (Participants) | 48
  4-weeks | 1.44 (0.94)
  8-weeks: number analyzed (Participants) | 44
  8-weeks | 1.23 (0.90)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .010, t-test, 2 sided; Slope = -0.04, Standard Error of Mean 0.02

3. Primary Outcome: Traumatic Stress - Hyperarousal Subscale
Description: as for outcome 2
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 1.61 (1.03)
  4-weeks: number analyzed (Participants) | 48
  4-weeks | 1.53 (1.04)
  8-weeks: number analyzed (Participants) | 44
  8-weeks | 1.31 (1.01)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .160, t-test, 2 sided; Slope = -0.02, Standard Error of Mean 0.02

4. Primary Outcome: Grief Intensity - Reality Subscale
Description: The Perinatal Grief Intensity Scale is 12 items that asks about an individuals' experiences with perinatal loss. Items are on a four-point scale from strongly disagree (1) to strongly agree (4). Three mean scale scores are computed including reality (5 items), congruence (4 items), and ability to confront others (2 items). Scores can range from 1 to 4 and higher scores indicate greater levels of grief intensity.
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 3.39 (0.57)
  4-weeks: number analyzed (Participants) | 48
  4-weeks | 3.41 (0.59)
  8-weeks: number analyzed (Participants) | 44
  8-weeks | 3.51 (0.60)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .167, t-test, 2 sided; Slope = 0.01, Standard Error of Mean 0.01

5. Primary Outcome: Grief Intensity - Congruence Subscale
Description: as for outcome 4
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 2.48 (0.60)
  4-weeks | 2.59 (0.59)
  8-weeks | 2.66 (0.58)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .012, t-test, 2 sided; Slope = 0.02, Standard Error of Mean 0.01

6. Primary Outcome: Grief Intensity - Ability to Confront Others Subscale
Description: as for outcome 4
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 2.61 (0.89)
  4-weeks | 2.71 (0.73)
  8-weeks | 2.55 (0.80)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .347, t-test, 2 sided; Slope = -0.01, Standard Error of Mean 0.01

7. Primary Outcome: Grief Management Self-efficacy
Description: Three items that rate the bereaved parents' confidence in their ability to cope with grief, use knowledge of mindfulness skills to cope, and engage in positive behaviors to help coping. Scores are on a six-point scale (1 to 6) with a mean total score that ranges from 1 to 6. Higher scores indicate greater self-efficacy.
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 4.26 (0.94)
  4-weeks | 4.63 (0.91)
  8-weeks | 4.66 (1.00)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .007, t-test, 2 sided; Slope = 0.05, Standard Error of Mean 0.02

8. Primary Outcome: Negative Attitudes on Personal Grief
Description: 6 items of experiences of care at the time of loss and follow-up appointments after loss. Responses on a 4-point scale from 1 (strongly disagree) to 4 (strongly agree) to indicate level of agreement. A means score was computed and could range from 1 to 4. Higher scores indicate more negative experiences.
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 3.88 (1.33)
  4-weeks: number analyzed (Participants) | 48
  4-weeks | 3.59 (1.22)
  8-weeks: number analyzed (Participants) | 44
  8-weeks | 3.21 (1.19)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .001, t-test, 2 sided; Slope = -0.08, Standard Error of Mean 0.02

9. Primary Outcome: Difficulties in Emotional Regulation - Nonacceptance of Emotional Response Subscale
Description: 11 items from the Difficulties in Emotional Regulation Scale (DERS) were assessed using a response option that ranged from 1 (almost never) to 5 (almost always). Two mean scale scores were computed including nonacceptance of emotional response (6 items) and lack of emotional awareness (5 items). Scale score could range from 1 to 5 with higher scores indicating greater difficulty regulating emotions.
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 2.25 (1.19)
  4 weeks: number analyzed (Participants) | 48
  4 weeks | 2.35 (0.93)
  8 weeks: number analyzed (Participants) | 44
  8 weeks | 2.08 (0.95)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .403, t-test, 2 sided; Slope = -0.02, Standard Error of Mean 0.02

10. Primary Outcome: Difficulties in Emotional Regulation - Lack of Emotional Response Subscale
Description: as for outcome 9
Time Frame: Baseline (immediately following loss), 4 weeks and 8 weeks post loss
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 52
units on a scale
  Pretest | 2.32 (0.77)
  4-weeks: number analyzed (Participants) | 48
  4-weeks | 2.38 (0.85)
  8-weeks: number analyzed (Participants) | 44
  8-weeks | 2.20 (0.79)
Statistical Analysis 1: Comparison: PeriGrief; Test type: Equivalence — Whether change in linear slope from pretest through the 8-week follow-up is equivalent to zero (null hypothesis); p = .194, t-test, 2 sided; Slope = -.02, Standard Error of Mean 0.01

11. Primary Outcome: Usability
Description: The System Usability Scale is commonly used 10-item scale that measures subjective perceptions of usability on a 5-point Likert-scale. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Higher scores indicate the technology is more usable.
Time Frame: Post-Treatment (8 weeks post loss)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 44
units on a scale | 74.4 (13.5)

12. Primary Outcome: Acceptability
Description: Developed as part of the current study, 7 items were designed to measure the degree, on a 5-point Likert-type scale (1 = strongly or somewhat disagree, 5 = strongly or somewhat agree) to which parents found the program helpful, acceptable, and suited to their needs. A mean score was computed across all items and could range from 1 to 5. Higher scores indicate greater acceptability.
Time Frame: Post-Treatment (8 weeks post loss)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PeriGrief
Number analyzed (Participants) | 45
units on a scale | 2.88 (0.29)

13. Primary Outcome: Program Use - Days Using the Program
Description: Program metrics on the backend of the program were used to track the total number of days the program was used.
Time Frame: Access to the program through through the study completion which was on average 2-months.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PeriGrief
Number analyzed (Participants) | 41
days | 21.40 (23.39)

14. Primary Outcome: Program Use - Modules Completed
Description: Program metrics on the backend of the program were used to track the the total number of modules completed out of the 6 modules.
Time Frame: Access to the program through through the study completion which was on average 2-months.
Measure: Count of Participants; unit: Participants
Arm/Group | PeriGrief
Number analyzed (Participants) | 41
Participants
  Did not complete any modules | 4
  Completed one module | 10
  Completed two modules | 9
  Completed three modules | 6
  Completed four modules | 1
  Completed five modules | 3
  Completed all six modules | 8

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from completion of consent form through the final 8-week assessment period.
Arm/Group | PeriGrief
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05318287/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05318287/ICF_001.pdf